CLINICAL TRIAL: NCT05564546
Title: Impact of Hydrogen Sulfide on Lung Health: Study of Chronic Exposure of the Population Living on the Atlantic Coast and on the Caribbean Coast, in Martinique, During the Stranding Period and Outside the Stranding Period of Sargassum Seaweeds
Brief Title: Study of Chronic Exposure of the Population Living on the Atlantic Coast and on the Caribbean Coast, in Martinique, During the Stranding Period and Outside the Stranding Period of Sargassum Seaweeds
Acronym: SÉSAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22_RIPH2-04; 2022-A01382-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2022-09-13; First posted 2022-10-03 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Ventilatory Disorders
Keywords: sargassum seaweed; exposure to H2S; pulmonary effects; H2S poisoning; fractional exhaled nitric oxide; spirometry
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: This is a prospective, longitudinal study, of exposed/non-exposed type, descriptive, comparative and monocentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People exposed to sargassum seaweed stranding (Experimental): Participant living on the Atlantic coast of Martinique island (hit by the strandings), close (less than 300 meters) to sargassum seaweed stranding areas: exposed group (85 subjects).
  Participants will be examined directly at their place of residence.
  Participants will be examinated two times:
  * at Visit 1 - Day 0 during the strandings period,
  * at Visit 2 - M+6 months (+/-1 month) after the end of the strandings.
  Interventions: Procedure: FeNO (fractional exhaled nitric oxide); Procedure: Spirometry; Other: Physical examination; Other: Interrogation
- People not exposed to sargassum seaweed stranding (Active Comparator): Participant living on the Caribbean coast of Martinique island (not hit by the strandings): unexposed group (85 subjects).
  Participants will be examined directly at their place of residence.
  Participants will be examinated two times:
  * at Visit 1 - Day 0 during the strandings period,
  * at Visit 2 - M+6 months (+/-1 month) after the end of the strandings.
  Interventions: Procedure: FeNO (fractional exhaled nitric oxide); Procedure: Spirometry; Other: Physical examination; Other: Interrogation

INTERVENTIONS:
Procedure: FeNO (fractional exhaled nitric oxide) — FeNO measurement is a marker of airway inflammation. It is a non-invasive examination for the patient, easy to perform for healthcare personnel, the measurement of NO in exhaled air is one of the only non-invasive and reproducible examinations allowing the detection of inflammation airways.
  The FeNO will be measured by an electrochemical NO analyzer of the NiOx Vero type (Circassia, The Surgical Company) and expressed in particles per billion (ppb). The objective and reproducible measurement of NO production by the bronchial mucosa is a reflection of the degree of airway inflammation. The measurement of exhaled NO is part of diagnostic health technologies aimed at quantifying airway inflammation, especially in asthmatic patients.
  FeNO is considered normal for values of 16-25 ppb. A FeNO value > 25 ppb will be a reason for consultation at the Martinique Hospital for additional assessment.
Procedure: Spirometry — Spirometry tests will assess lung function. It is a safe and painless test to measure lung volumes and expiratory flows.
  Ventilatory function is assessed by simple spirometry parameters such as forced expiratory volume in the first second (FEV1, in litres), vital capacity (CV, in litres), and the FEV1/CV ratio.
  The results of the spirometry will be compared with the theoretical or predicted values calculated according to age, sex, height.The FEV1/CV ratio as a percentage is an indicator of the level of bronchial obstruction.
  Spirometry is considered normal for CV values ≥80% and FEV1/FVC ≥0.70 of the predicted value. A value of CV <80% or FEV <80% of the predicted value will be a reason for consultation at the Martinique hospital for additional assessment.
Other: Physical examination — A pulmonary clinical examination will be carried out by the investigator, including:
  * Cough,
  * Sputum,
  * Vesicular murmur (MV),
  * Added noises (BSA),
  * Vocal vibrations (VV),
  * Tympanism,
  * Dullness,
  * Signs of acute respiratory distress (ARD),
  * …
Other: Interrogation — Participants will undergo an interview with the medical team to collect the following information in particular:
  Age, size, sex, medical history, smoking status, current treatments, potential symptoms, date of first symptoms, clinical manifestations experienced (respiratory, digestive, neurological, cardiac, psychiatric, visual, skin disorders, etc.) place of residence, concentration H2S in ppm on the site, presence of sand mist in the environment, etc.

SUMMARY:
Sargassum are pelagic brown sea algae. Two species grow on the surface of the ocean and drift freely with ocean currents in the form of slicks: the pelagic Sargassum fluitans and Sargassum natans.

Since 2011, massive strandings of Sargassum seaweed in the French West Indies are to be deplored. In recent years, strandings have increased. In Martinique, sargassum stranding occurs mainly on the Atlantic coast. The duration of stranding from one year to another is variable, but the period during which the stranding is maximum is between April and October.

The accumulation of strandings causes the compaction of algae and limits access to oxygen, which leads to anaerobic degradation which quickly results in the release of various gases, in particular hydrogen sulphide (H2S).

Acute H2S poisoning is well characterized clinically according to exposure (cutaneous, respiratory, ophthalmological, digestive, neurological symptoms, etc.). On the other hand, there are very few data available on the clinical effects of prolonged, repeated exposure and most often at low doses.

Among the toxic effects for which there are still uncertainties regarding long-term exposure to H2S are lung function, measured by spirometry, and airway inflammation, appreciable by measurement of FeNO (fractional exhaled nitric oxide).

The investigators consider it relevant to focus on the clinical and biological characteristics of the population exposed to sargassum in Martinique, in the field, assuming that exposure to sargassum H2S causes pulmonary effects measurable by spirometry and by FeNO, during the stranding period and outside this period.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant (age greater than or equal to 18),
* Participant living on the Atlantic coast in Martinique, close (less than 300 meters) to sargassum seaweed stranding areas (exposed group),
* Participant living on the Caribbean coast, in Martinique (unexposed group),
* Participant having been informed of the research,
* Participant having given his free, informed and express consent,
* Participant affiliated to a social security scheme.

Exclusion Criteria:

* Minor Participant,
* Participant with a known respiratory or cardiac pathology,
* Participant with a cognitive state that does not allow him to answer the questionnaire,
* Participant who refused to participate in the study,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Compare the expired fractions of nitric oxide between people exposed and not exposed to toxic gases from sargassum in Martinique | 6 months
  The primary endpoint of the study will be FeNO (exhaled fraction of nitric oxide). FeNO measurement is a marker of airway inflammation. This is a test used routinely for the non-invasive detection and quantification of bronchial inflammation.
  FeNO is considered normal for values of 16-25 ppb. A FeNO value > 25 ppb will be a reason for consultation at the Martinique Hospital for additional assessment.

SECONDARY OUTCOMES:
Compare the pulmonary effects (spirometric) related to the emission of toxic gases from Sargassum between people exposed and those not exposed to Sargassum in Martinique. | 6 months
  The pulmonary effects related to the emission of toxic gases from Sargassum between exposed and non-exposed people will be compared based on the slow and forced spirometry measurements.
  Spirometry tests will assess lung function. It is a safe and painless test to measure lung volumes and expiratory flows.
  Ventilatory function is assessed by simple spirometry parameters such as forced expiratory volume in the first second (FEV1, in litres), vital capacity (CV, in litres), and the FEV1/CV ratio.
  The results of the spirometry will be compared with the theoretical or predicted values calculated according to age, sex, height.The FEV1/CV ratio as a percentage is an indicator of the level of bronchial obstruction.
  Spirometry is considered normal for CV values ≥80% and FEV1/FVC ≥0.70 of the predicted value. A value of CV <80% or FEV <80% of the predicted value will be a reason for consultation at the Martinique hospital for additional assessment.
Compare the pulmonary effects (clinical) related to the emission of toxic gases from Sargassum between people exposed and those not exposed to Sargassum in Martinique. | 6 month
  The pulmonary effects related to the emission of toxic gases from Sargassum between exposed and non-exposed people will be compared based on the clinical examination results.
  A pulmonary clinical examination will be carried out by the investigator, including:
  Cough, Sputum, Vesicular murmur (MV), Added noises (BSA), Vocal vibrations (VV), Tympanism, Dullness, Signs of acute respiratory distress (ARD), Respiratory rate, SpO2…
  In addition, participants will undergo an interview with the medical team to collect the following information in particular:
  Age, size, sex, medical history, smoking status, current treatments, potential symptoms, date of first symptoms, clinical manifestations experienced (respiratory, digestive, neurological, cardiac, psychiatric, visual, skin disorders, etc.) place of residence, concentration H2S in ppm on the site, presence of sand mist in the environment, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, France